CLINICAL TRIAL: NCT05793944
Title: Teaching by Texting to Promote Health Behaviours in Pregnancy
Brief Title: SmartMom: Teaching by Texting to Promote Health Behaviours in Pregnancy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Patricia Janssen, Professor, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: H22-00603
Record Dates: First submitted 2023-01-30; First posted 2023-03-31 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Pregnancy
Keywords: prenatal education; perinatal outcomes; text messaging; mobile health; mental health; health behaviour
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention: SmartMom messaging (Active Comparator): Participants receive three text messages per week with evidence-based information to promote healthy behaviours during pregnancy.
  Interventions: Behavioral: SmartMom text messaging
- Control messaging (Placebo Comparator): Participants receive one text message per week with general information about pregnancy but not about making healthy choices.
  Interventions: Behavioral: Control text messaging

INTERVENTIONS:
Behavioral: SmartMom text messaging — SmartMom is a mobile health program delivered via text messaging that guides participants through each week of pregnancy. Participants receive three messages per week with links to content focused on improving knowledge, providing information about prenatal assessments and screening, and encouraging the adoption of behaviours to support healthy pregnancy and physiologic birth. Messages are consistent with current professional guidelines and peer reviewed prenatal education curricula. SmartMom provides optional supplemental streams for individuals who wish to have additional messages addressing topics such as reducing use of tobacco, alcohol or illicit drugs, depression, obesity, and maternal age over 35.
  Arms: Intervention: SmartMom messaging
Behavioral: Control text messaging — Control arm participants will receive weekly text messages with accurate, general-interest information about pregnancy and about progress of the trial. Content is not geared to decision-making during pregnancy that may affect health outcomes.
  Arms: Control messaging

SUMMARY:
The goal of this randomized clinical trial is to evaluate the effectiveness of SmartMom, a text messaging-based mobile health program for prenatal education. The main questions are to determine if healthy pregnant people receiving SmartMom messages that promote health behaviours in pregnancy versus messages that don't provoke behaviour change have improvement in:

1. knowledge about healthy pregnancy and birth
2. standardized measures of depression, anxiety, and fear of childbirth
3. adoption of positive health behaviours in pregnancy
4. maternal, fetal, and newborn outcomes

Participants in the intervention group will receive three evidence-based text messages per week, plus optional supplemental messages on topics relevant to them, throughout pregnancy.

The control group will receive general interest messages on pregnancy-related topics that are not promoting behaviour change.

ELIGIBILITY:
Inclusion Criteria:

* pregnant person
* at 15 weeks gestation or earlier
* singleton pregnancy
* can read and understand English at grade 8 level and comfortable completing online surveys
* live in Canada (excluding British Columbia where SmartMom has been piloted)

Exclusion Criteria:

* health conditions existing prior to pregnancy that require individualized care (e.g. hypertension, cardiac disease, diabetes)
* previously had a baby with the SmartMom program

Min Age: 15 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 3078 (Estimated)
Dates: Start 2023-11-10 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Change in weight during pregnancy | Enrollment, 38 weeks gestation
  Rate of pregnancy weight gain in a range appropriate for pre-pregnancy BMI. These include self-reported data as well as data from provincial prenatal registries and the Canadian Hospital Discharge Database linked via personal health number, provided as part of the consenting procedure.
Attendance at prenatal care visits through pregnancy | 38 weeks gestation
  Rates of attendance at prenatal care appointments in adherence to Canadian guidelines. These include self-reported data as well as data from provincial prenatal registries and the Canadian Hospital Discharge Database linked via personal health number, provided as part of the consenting procedure.

SECONDARY OUTCOMES:
Changes in health knowledge through pregnancy | Enrollment, 38 weeks gestation
  Changes in health knowledge as measured by a 10-item knowledge test. Minimum score = 0, Maximum score = 10. Higher score indicates more knowledge i.e. more positive outcome.
Health literacy at end of pregnancy | 38 weeks gestation
  Health literacy as measured by self-report of i) information-seeking from local health and social services resources; ii) awareness of their choices regarding serum genetic screening; iii) awareness of their choices to have (yes/no) serum glucose screening.
Changes in fear of childbirth through pregnancy | Enrollment, 38 weeks gestational age
  Changes in fear of childbirth as measured by The Childbirth Fear Scale, an 11-item, self-reported measure.
  Minimum score = 6, Maximum score = 66. Lower score means less fear, i.e. a more positive outcome.
Changes in depression through pregnancy | Enrollment, 38 weeks gestational age
  Changes in depression as measured by the Edinburgh Postnatal Depression Scale. This is a 10-item, self-report screening tool for postnatal depression that is also valid for use during pregnancy.
  Minimum score = 0. zero, Maximum score = 30. Lower score means less depression, i.e. a more positive outcome.
Changes in anxiety through pregnancy | Enrollment, 38 weeks gestational age
  Changes in anxiety as measured by the standardized 33-item Pregnancy Specific Anxiety Tool (PSAT).
  Minimum score = 6, Maximum score = 24. Lower score means less anxiety, i.e. a more positive outcome.
Changes in use of tobacco, vaping, alcohol, or cannabis through pregnancy among users. | Enrollment, 38 weeks gestational age
  Among participants indicating that they are users of tobacco, vaping, alcohol, and/or cannabis at enrollment, change of use at the end of pregnancy will be measured by self-report.
  Report: proportion of users that stopped using per trial arm. Among users continuing to use: mean change in number of daily cigarettes, episodes of vaping, drinks per week, cannabis products per day or other specified use of recreational or prescription drugs used per day.
Rates of planned vaginal birth after cesarean | 38 weeks gestation
  Proportion of participants choosing to plan vaginal birth (VBAC) after a previous cesarean birth, among those deemed eligible by their caregivers.
  These include self-reported data as well as data from provincial prenatal registries and the Canadian Hospital Discharge Database linked via personal health number, provided as part of the consenting procedure.
Rates of exclusive breastfeeding at hospital discharge | 1 month post birth
  These include self-reported data as well as data from provincial prenatal registries and the Canadian Hospital Discharge Database linked via personal health number, provided as part of the consenting procedure.
Rates of adverse pregnancy outcomes as measured by gestational diabetes, stillbirth, preterm birth (<37 weeks gestation) and small for gestational age (SGA) status at birth. | 1 month post birth
  These include self-reported data as well as data from provincial prenatal registries and the Canadian Hospital Discharge Database linked via personal health number, provided as part of the consenting procedure.
Incremental costs per incidence of suboptimal weight gain and inadequate prenatal care avoided. | Throughout pregnancy (up to 42 weeks) and birth, including hospital admission in which birth took place (up to 7 days).
  Incremental costs per incidence of suboptimal weight gain and inadequate prenatal care avoided for the intervention group when compared to control group as an incremental cost-effectiveness ratio.

CONTACTS AND LOCATIONS:
Overall Officials: Patti Janssen, PhD, Principal Investigator — University of British Columbia
Locations (1):
- BC Children's Hospital Research Institute, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data will be available from the corresponding author upon reasonable request including a research proposal outlining how the data will be used and a certificate of ethical approval from an academic ethics review board.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: At completion of study enrollment for five years
Access Criteria: Available to academic researchers who have submitted a research protocol that has been approved by a university ethics board.

REFERENCES:
- [Background] Debessai Y, Costanian C, Roy M, El-Sayed M, Tamim H. Inadequate prenatal care use among Canadian mothers: findings from the Maternity Experiences Survey. J Perinatol. 2016 Jun;36(6):420-6. doi: 10.1038/jp.2015.218. Epub 2016 Jan 21. PMID 26796126
- [Background] Dzakpasu S, Fahey J, Kirby RS, Tough SC, Chalmers B, Heaman MI, Bartholomew S, Biringer A, Darling EK, Lee LS, McDonald SD. Contribution of prepregnancy body mass index and gestational weight gain to adverse neonatal outcomes: population attributable fractions for Canada. BMC Pregnancy Childbirth. 2015 Feb 5;15:21. doi: 10.1186/s12884-015-0452-0. PMID 25652811
- [Background] Ganer Herman H, Dekalo A, Jubran L, Schreiber L, Bar J, Kovo M. Obstetric outcomes and placental findings in gestational diabetes patients according to maternal prepregnancy weight and weight gain. J Matern Fetal Neonatal Med. 2019 May;32(10):1682-1687. doi: 10.1080/14767058.2017.1416078. Epub 2018 Feb 5. PMID 29402158
- [Background] Munro S, Hui A, Salmons V, Solomon C, Gemmell E, Torabi N, Janssen PA. SmartMom Text Messaging for Prenatal Education: A Qualitative Focus Group Study to Explore Canadian Women's Perceptions. JMIR Public Health Surveill. 2017 Feb 7;3(1):e7. doi: 10.2196/publichealth.6949. PMID 28174149
- [Background] van den Heuvel JF, Groenhof TK, Veerbeek JH, van Solinge WW, Lely AT, Franx A, Bekker MN. eHealth as the Next-Generation Perinatal Care: An Overview of the Literature. J Med Internet Res. 2018 Jun 5;20(6):e202. doi: 10.2196/jmir.9262. PMID 29871855
- [Derived] Ennis M, Renner RM, Morando-Stokoe C, James S, Janssen PA, Leckie S, Dunn S, Mazza D, Norman WV. Exploring Methods to Mitigate Fraud in Web-Based Surveys: Multicase Study Analysis. J Med Internet Res. 2025 Dec 1;27:e78671. doi: 10.2196/78671. PMID 41324984
- [Derived] Janssen P, Lecke S, Renner R, Zhang W, Vedam S, Norman WV, Bayrampour H, Tough S, Murray J, Muhajarine N, Dennis CL. Teaching by texting to promote positive health behaviours in pregnancy: a protocol for a randomised controlled trial of SmartMom. BMJ Open. 2024 Jan 18;14(1):e081730. doi: 10.1136/bmjopen-2023-081730. PMID 38238058